CLINICAL TRIAL: NCT03844581
Title: Effect of Interferential Electrical Stimulation on Pain Perception and Disability Level on Interstitial Cystitis
Acronym: IF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ghada Ebrahim El Refaye, assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CairoU6
Record Dates: First submitted 2019-02-15; First posted 2019-02-18 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Interstitial Cystitis
MeSH Terms: conditions — Cystitis, Interstitial | interventions — Electric Stimulation Therapy; propiverine

STUDY DESIGN:
Intervention Model Description: A total of 40 volunteers women with a diagnosis of interstitial cystitis. Their ages ranged from 25 to 40 years old; their body mass index was > 30 kg/m2 and were randomly assigned to a group (A) received interferential current at the lower abdomen, and also received traditional medicine or group (B) received traditional medicine for 8 successive weeks.
Who Masked: Participant, Investigator
Masking Description: Participants were assigned randomly used sealed envelope
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interferential current (Active Comparator): interferential current with a constant frequency of 100Hz for pain relief, then using rhythmic frequency of 1-100 Hz that help to disperse infiltration and adhesions for 8 successive weeks
  Interventions: Device: interferential current
- anticholinergics (Active Comparator): anticholinergics (propiverine hydrochloride 20 mg/once per day in the morning) for 8 successive weeks
  Interventions: Drug: Propiverine Hydrochloride

INTERVENTIONS:
Device: interferential current — Treatment was applied using four vacuum electrodes with wet sponge, two of them were put under the patient lumber region on a distance from lumber spinous process by five cm on each side and the other two were applied over the suprapubic region parallel to iliac crest.
  Arms: interferential current
Drug: Propiverine Hydrochloride — propiverine hydrochloride 20 mg/once per day in the morning
  Arms: anticholinergics

SUMMARY:
A total of 40 volunteers women with a diagnosis of interstitial cystitis. Their ages ranged from 25 to 40 years old; their body mass index was > 30 kg/m2 and were randomly assigned to a group (A) received interferential current at the lower abdomen, and also received traditional medicine or group (B) received traditional medicine for 8 successive weeks. Both of the groups received the treatment program for 8 successive weeks. Assessment of pain perception and disability level for all patients in both groups (A&B) were done through Visual analogue scale, O'Leary-Sant Symptom Index or Interstitial Cystitis Index (ICSI) and blood cortisol concentration were done before and after the treatment program.

DETAILED DESCRIPTION:
Forty volunteers women diagnosed clinically by gynecologist as painful bladder syndrome were participated in this study. They were selected randomly from the gynecological outpatient clinic, at Al-Zahra Universal Hospital, Al Azhar University, their ages ranged from 25 to 40 years and their body mass index was > 30 kg/m2. All participants complain from suprapubic pain related to bladder filling, accompanied by other symptoms such as increased daytime and night-time frequency. Exclusion criteria of the study were as follows: Participant who had acute viral disease, acute tuberculosis and mental disorders, benign or malignant tumors of the pelvic region, Participant who had active endometriosis or having artificial pacemaker or cardiac arrhythmia, Participant who had sensory disturbances.

Participants were assigned randomly used sealed envelope into two groups (A&B) equally in number. Group (A): Consisted of twenty patients suffering from painful bladder syndrome. They received interferential current at the lower abdomen, and also received traditional medicine (they were administered anticholinergics (propiverine hydrochloride 20 mg/once per day in the morning) for 8 successive weeks. Group (B): Consisted of twenty patients suffering from painful bladder syndrome. They received traditional medicine (they were administered anticholinergics (propiverine hydrochloride 20 mg/once per day in the morning) for 8 successive weeks

ELIGIBILITY:
Inclusion Criteria:

* their ages ranged from 25 to 40 years.
* their body mass index was > 30 kg/m2

Exclusion Criteria:

* Participant who had acute viral disease.
* acute tuberculosis
* mental disorders.
* benign or malignant tumors of the pelvic region

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-02-13 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale | 8 weeks
  pain was assessed by the visual analogue scale to all participants in both two groups (A, B)

SECONDARY OUTCOMES:
O'Leary-Sant Symptom Index or Interstitial Cystitis Index (ICSI) | 8 weeks
  It is useful in assessing baseline symptoms (including pain, frequency, nocturia and impact on activities) and effectiveness of treatments. The Interstitial Cystitis Problem Index (ICPI) documents symptom bother.
Plasma cortisol concentration | 8 weeks
  5 ml of venous blood were drawn from the patient at the morning (at 9 am), put into a tube to measures the level of cortisol in the blood.

CONTACTS AND LOCATIONS:
Overall Officials: ghada eb elrefaye, professor, Principal Investigator — Department of Physical Therapy for Women's Health, Faculty of Physical therapy, Cairo University, Egypt.
Locations (2):
- Egypt (2):
  - Faculty of physical therapy- Cairo University, Giza, Dokki
  - Al Azhar University, Cairo

IPD SHARING:
Plan to Share IPD: Undecided